CLINICAL TRIAL: NCT00599131
Title: A Phase II Organ Preservation Trial Using Cetuximab and Radiation Therapy in Advanced Laryngeal Cancer Patients Who Have Responded to One Cycle of Induction Chemotherapy With Taxotere, Cisplatin, 5-Fluorouracil (TPF), and Cetuximab
Brief Title: Cetuximab and Radiation Therapy in Laryngeal Cancer Patients Who Have Responded to One Cycle of Chemotherapy (SPORE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued prematurely due to early stopping rules.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.029; HUM 11350 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-12; First posted 2008-01-23 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Cancer of Larynx
Keywords: Cancer of Larynx
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Cisplatin; Cetuximab; Fluorouracil; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy/Radiation/Surgery (Experimental): Patients will undergo induction chemotherapy with (TPF): Docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 on day 1, and 5-FU 750 mg/m2 days 1-4.
  On day 20 patients will receive a single dose of cetuximab (C-225) 400 mg/m2.
  Depending upon disease response, patients will undergo salvage laryngectomy followed by radiation therapy and chemotherapy.
  Interventions: Drug: Cisplatin; Drug: Cetuximab; Drug: 5-Fluorouracil; Drug: Docetaxel

INTERVENTIONS:
Drug: Cisplatin — 1. Day 1: 100 mg/m2, administered as an i.v. infusion will run over one hour. 2. Day #23: Subjects with a < 50% response (NR) to induction chemotherapy will undergo salvage laryngectomy followed by RT. Cisplatin will be added to radiation for patients whose surgical pathology reveals high-risk features (i.e. extracapsular spread, > 2 positive lymph nodes, perineural invasion, or positive margins). Cisplatin will either be dosed a 100 mg/m2 every 21 days or 40 mg/m2 weekly at the discretion of the prescribing physician.
  Other Names: Platinol®-AQ
Drug: Cetuximab — 1. Cetuximab will be administered at 400 mg/m2 on Day 20 (2 hour administration). 2. Cetuximab will be administered in combination with radiation therapy to those subjects who had a Partial or Complete response after the first cycle of the chemotherapy regimen is administered. The dosage for these administrations is 250 mg/m2 over sixty minutes and it will be administered for six weeks.
  Other Names: C-225; Erbitux®
Drug: 5-Fluorouracil — 5-FU will be administered 750 mg/m2 in 0.9% normal saline as a 24-hour continuous infusion, days #1-4.
  Other Names: Adrucil®; Carac™; Efudex®; Fluoroplex®; 5-FU; FU
Drug: Docetaxel — 75 mg/m2 by I.V. over one hour on Day # 1 only
  Other Names: Taxotere®

SUMMARY:
The purpose of this study is to learn how to identify early which patients will respond to chemotherapy plus radiation therapy in order to reduce the number of subjects who require surgery (followed by radiation therapy).

DETAILED DESCRIPTION:
In this study one cycle of chemotherapy will be administered and then those subjects who respond well to that cycle will be started on radiation therapy along with chemotherapy and those that don't respond well to the initial cycle of chemotherapy, will undergo a total laryngectomy (surgery to remove the voice box) followed by radiation therapy. The initial cycle of chemotherapy consists of the drugs Taxotere, Cisplatin, and 5-Fluorouracil (this combination is known as TPF). Then on Day 20 of the study, the subjects will be administered another chemotherapy agent called cetuximab (a.k.a. C-225). It will then be determined if the patient's response to the chemotherapy was favorable by examining the patient's tumor with an endoscopy. If the response is determined to be good, then the patient will continue with a chemotherapy regimen with the addition of radiation therapy combination. If the patient's response to the chemotherapy is determined to be less than favorable, then the patient will be advised to undergo salvage surgery (a.k.a. laryngectomy) to remove their voice box and then undergo radiation therapy treatment. Additionally, tumor tissue samples and blood will be studied to see if there are special molecular markers that help predict when a tumor will respond to chemotherapy and radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed, previously untreated, resectable, squamous cell carcinoma of the larynx.
* Disease must be Stage III or IV.
* Tumor must be potentially surgically resectable and curable with conventional surgery and radiation therapy.
* Patients must undergo pre-treatment endoscopic tumor staging and CT scanning.
* ECOG Performance status 0-2
* Pre-treatment laboratory criteria:
* WBC > or = to 3500/ul, granulocyte > or = to 1500/ul.
* Platelet count > or equal to 100,000/ul.
* Calculated or measured creatinine clearance > or = to 60 cc/min.
* Total Bilirubin < or = to 1.5 X ULN.
* AST and ALT < or = to 2.5 X ULN.
* Patients must give documented informed consent to participate in this study.

Exclusion Criteria:

* Prior head and neck malignancy or history of other prior non-head and neck malignancy within the past 3 years.
* Prior head and neck radiation or prior chemotherapy.
* Documented evidence of distant metastases.
* Active infection.
* Pregnancy or lactation. Patients must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Any medical or psychiatric illness which in the opinion of the principal investigator would compromise the patients ability to tolerate this treatment.
* Patients residing in prison.
* Age < 18 years.
* Patients with psychiatric/social situations that would limit compliance with study requirements are not eligible.
* Patients with prior radiation to the head and neck.
* Patients with prior anti-epidermal growth-factor receptor antibody therapy or therapy with a tyrosine-kinase inhibitor.
* Patients with Grade > 2 peripheral neuropathy.
* Any history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P. Worden, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy/Radiation/Surgery
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 54 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Histologic Complete Response
Description: The proportion of patients treated with radiation+cetuximab achieving histologic CR will be estimated, along with 95% exact confidence intervals. Histologic Complete Response (CR) will be defined as primary tumors exhibiting a clinical CR or at least a 90% PR (Partial Response) along with a negative post-treatment biopsy.
Time Frame: 3 years
Population: The study was discontinued prematurely due to an early stopping rule. No participants were assessed for the primary outcome because an insufficient number of patients were recruited.
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: The Difference, From Baseline, in EGFR, for Tumor Biopsies Taken After the Administration of Cetuximab Following TPF.
Description: To determine tumor EGFR degradation, as well as other markers of down-stream EGFR inhibition, observed in tumor biopsies taken shortly after the administration of cetuximab following TPF, compared with pre-treatment biopsies.
Time Frame: Day 23
Population: The study was discontinued prematurely due to an early stopping rule. No participants were assessed because an insufficient number of patients were recruited.
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 0

3. Secondary Outcome: The Change in Overall Quality of Life Score During Radiation Therapy and at 6, 12, and 24 Months Post Treatment.
Description: To evaluate the quality of life (QOL).
Time Frame: 24 months
Population: as for outcome 2
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival Time
Description: To determine the overall survival rates compared to the overall survival rates of historical controls.
Time Frame: 3 years
Population: as for outcome 2
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 0

5. Secondary Outcome: The Number of Patients That Experience Grade 3 and 4 Mucositis or Dysphagia
Description: To determine and compare toxicities, most notably mucositis and dysphagia, in patients on this treatment regimen as compared to historical controls.
Time Frame: 3 years.
Population: as for outcome 2
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy/Radiation/Surgery
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy/Radiation/Surgery (N=4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Colitis, Infection (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infection with Grade 3-4 Neutrophils (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy/Radiation/Surgery (N=4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (2)
Weight loss (General disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 4 (4)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 4 (8)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam), Oral Cavity (Investigations) | 3 (9)
Mucositis/stomatitis (clinical exam), Pharynx (Investigations) | 3 (7)
Mucositis/stomatitis (functional/symptomatic), Oral Cavity (Gastrointestinal disorders) | 2 (5)
Mucositis/stomatitis (functional/symptomatic), Pharynx (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Skin Infection with Grade 3 or 4 neutrophils (Skin and subcutaneous tissue disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Foreign Body) (Infections and infestations) | 1 (1)
Infection (Upper Aerodigestive, NOS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Upper Airway, NOS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection with unknown ANC (Upper Aerodigestive) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle weakness, Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (3)
Confusion (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 2 (2)
Ocular/Visual - Other (Specify) (Eye disorders) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (2)
Head Pain (Nervous system disorders) | 2 (2)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Throat Pain (Gastrointestinal disorders) | 3 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fistula, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sexual/Reproductive Function - Other (Specify) (Reproductive system and breast disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (12)

LIMITATIONS AND CAVEATS:
The study was discontinued prematurely due to an early stopping rule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No